CLINICAL TRIAL: NCT06200233
Title: A Phase II, Open-label, Single-arm, Multi-center Clinical Trial of Rivoceranib in Patients With Metastatic Thymic Epithelial Tumor
Brief Title: Rivoceranib in Patients With Metastatic Thymic Epithelial Tumor
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, M.D. Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-09-121
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Thymic Epithelial Tumor
MeSH Terms: conditions — Thymic epithelial tumor | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Rivoceranib 700 mg once daily by mouth. Rivoceranib should be given at the same time each day, with or without meals. Swallow the tablet whole. Do not chew, crush, or split the tablet.
  Receive study medication until there is evidence of disease progression, intolerable toxicity, withdrawal of consent by the patient, or in the judgment of the principal investigator that the study cannot continue due to inability to administer.
  Tumor response will be assessed according to RECIST v1.1 criteria based on imaging studies (CT or MRI) measured every 8 weeks (±1 week) from C1D1 through 12 months and every 12 weeks (±1 week) after 12 months.
  Interventions: Drug: Rivoceranib

INTERVENTIONS:
Drug: Rivoceranib — 700mg once daily

SUMMARY:
PURPOSE: To evaluate the efficacy and safety of Rivoceranib in patients with metastatic thymic epithelial tumors who developed resistance on first-line therapy.

Study Design: Patients with histologically confirmed metastatic thymic epithelial tumors who meet the inclusion/exclusion criteria will be enrolled in this study. In Stage 1, 18 subjects will be enrolled to receive study medication. If a tumor response is observed in at least 5 of these subjects, the study will proceed to Stage 2 to enroll the remaining subjects, or the study will be stopped early due to lack of clinical benefit of the investigational product. The trial will be considered clinically valid if a response is observed in 11 or more subjects out of a total of 33 subjects. Investigational product(Rivoceraniv 700 mg) will be administered until disease progression, development of intolerable adverse events, death, withdrawal of consent by the subject, or when, in the opinion of the principal investigator, it is inappropriate or impossible to continue the study. Imaging studies (CT or MRI) will be performed every 8 weeks (+,- 1 week) for C1D1 through 12 months and every 12 weeks (+,- 1 week) after 12 months, and the results will be used to assess tumor response according to RECIST v1.1 criteria. Safety will be assessed at C1D1, C1D7, and each scheduled visit thereafter.

DETAILED DESCRIPTION:
Thymic epithelial tumors (TET) are tumors of the thymus gland, which plays a pivotal role in adaptive immunity, and are classified as thymoma, thymic carcinoma, and thymic neuroendocrine tumor. Although it is the most common neoplasm of the anterior mediastinum, it is a rare cancer with an incidence of 0.15 cases per 100,000 people per year in the United States and 1.7 cases per 1,000,000 people per year in Europe. For surgically inoperable thymic epithelial tumors, first-line treatment is based on cytotoxic anticancer drugs. In this case, combinations such as Paclitaxel/Carboplatin or Cyclophosphamide, Adriamycin, Cisplatin (CAP) are mainly used as first-line treatment, but their therapeutic effect is still limited to less than 40%, and they also have very high toxicity. In the event of resistance to first-line therapy, there are a number of treatment options available, including Sunitinib, Pemetrexed, Everolimus, Paclitaxel, Gemcitabine based regimens, Lenvatinib, and Pembrolizumab. Lenvatinib, a representative agent with a similar mechanism of action to rivoceranib, has also shown excellent clinical results in thymic epithelial tumors. Lenvatinib, which targets various kinases in addition to the Vascular Endothelial Growth Factor Receptor (VEGFR), was used in a total of 42 patients, resulting in a partial response in 38% of patients and stable disease in 57% of patients. Rivoceranib is a selective inhibitor of VEGFR-2 and is currently approved and marketed in China for the treatment of gastric and liver cancer. Rivoceranib has similar targets to Lenvatinib and Sunitinib, and this study is expected to show clinical benefits when used in thymic epithelial tumors (TET), providing additional treatment opportunities for patients in the absence of targeted therapies currently covered by domestic insurance in the second-line setting.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older at the time of signing informed consent
2. Subjects with histologically confirmed metastatic thymic epithelial tumor
3. Have at least one measurable target lesion for evaluation according to RECIST v1.1 criteria
4. Patients who are not candidates for surgery and require consolidation chemotherapy
5. Radiologic progression of disease after first-line standard therapy
6. ECOG performance status of 0 or 1
7. Life expectancy greater than 3 months
8. Patients with adequate bone marrow and organ function [Bone marrow function]

   * Neutrophils (ANC) > 1,500/mm3
   * Platelets > 100,000/mm3
   * Hemoglobin > 9 g/dL [Liver function]
   * Total bilirubin ≤ 1.5 x upper limit of normal (if liver metastases are present, up to 3 x upper limit of normal is allowed)
   * AST, ALT ≤ 3 x upper limit of normal (if liver metastases are present, up to 5 x upper limit of normal is allowed) [Renal function]
   * Creatinine clearance > 50 mL/min (Cockcroft-Gault equation)
9. Subjects who have voluntarily decided to participate in this study and have given written informed consent and are able to participate in all periods of the study.

Exclusion Criteria:

1. Patients with more than 22 concurrent tumors and/or other active malignancies requiring systemic treatment within the last 22 years at the time of the first dose of investigational drug (however, patients may participate in the study if the principal investigator determines that the previous malignancy has been treated and no further treatment is required).
2. Patients treated with a previous anti-angiogenic agent (ex. Sunitinib, bevacizumab etc)
3. Patients with difficult to control central nervous system metastases
4. Those with spinal cord compression, leptomeningeal carcinomatosis
5. Patients with uncontrolled systemic disease, including uncontrolled hypertension, active bleeding, or active infection.

   However, individuals with the following hepatitis B/C infections may be enrolled
   * Hepatitis B surface antigen (HBsAg) positive, with an ALT in the normal range and HBV DNA <2,000 IU/ml, and taking antiviral therapy to prevent hepatitis reactivation may be enrolled.
   * HBs Ag negative, hepatitis B core antibody (IgG anti-HBc) positive, and HBV DNA below the lower limit of quantification may be enrolled.
   * Anti-HCV Ab positive individuals can be enrolled if HCV RNA is the lower limit of quantification.
6. Unresolved toxicities from prior therapy greater than or equal to grade 1 based on CTCAE version 5.0.
7. Received extensive radiotherapy within the last 2 weeks, or received localized radiotherapy or gamma knife surgery with a limited scope of radiotherapy for palliative purposes within the last 1 week.
8. Unable to swallow investigational medication due to intractable nausea and vomiting or chronic gastrointestinal disease.
9. Participation in another interventional clinical trial within 30 days of screening
10. Pregnant or lactating women
11. Unwilling to agree to use a medically acceptable method of contraception from the first dose of investigational drug until 1 month after the last dose.

    * Female patients of childbearing potential who are sexually active and their partners must agree to use adequate medically acceptable contraception for the duration of the study and for 1 month after the last dose.
    * Male patients who have not undergone a vasectomy must agree to use adequate contraception and are prohibited from providing sperm until 1 month after the last dose of study medication.

      * Adequate contraception includes: hormonal contraceptives (subcutaneous fat, injections, oral contraceptives, etc.), intrauterine devices (IUD, intrauterine device or IUS, intrauterine system), sterilization of you or your partner (vasectomy, tubal ligation, etc.).
12. Failure to provide 20 unstained slides (if additional biopsies are not available from the patient, participation in the study may be possible after discussion with the study coordinator).
13. Those who are inappropriate to participate in the study for other reasons (e.g., ethically or because it may affect the outcome of the study) as judged by the principal investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) Objective response rate(ORR) | 6 month after completion of enrollment

SECONDARY OUTCOMES:
Progression-free survival(PFS) | up to 30 months
Disease control rate(DCR) | up to 30 months
Duration of response(DOR) | up to 30 months

OTHER OUTCOMES:
Exploratory biomarker analysis | up to 30 months
  Genomic analysis (whole transcriptome sequencing) - Circulating tumor DNA
Exploratory biomarker analysis | up to 30 months
  Tissue slide - Whole transcriptome sequencing, Whole exome sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea